CLINICAL TRIAL: NCT03580473
Title: Phase II, National, Multicenter, Randomized, Double Blind Clinical Trial, to Evaluate the Efficacy and Safety of Saturno IIB Association on the Control of Ocular Inflammation Post-phacoemulsification
Brief Title: Efficacy and Safety of Saturno IIB Association on the Control of Ocular Inflammation Post-phacoemulsification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMS0118-SATURNO II
Record Dates: First submitted 2018-05-23; First posted 2018-07-09 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Ocular Inflammation; Cataract
MeSH Terms: conditions — Cataract | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SATURNO II (Experimental): 1 drop, 4 times a day, in the eye to be operated, 1 day before surgery until 15 days after surgery
  Interventions: Drug: SATURNO II association
- Vigadexa® (Active Comparator): 1 drop, 4 times a day, in the eye to be operated, 1 day before surgery until 15 days after surgery
  Interventions: Drug: Vigadexa®

INTERVENTIONS:
Drug: SATURNO II association — opthalmic solution, 4 times a day
  Other Names: Legrand association
  Arms: SATURNO II
Drug: Vigadexa® — opthalmic solution, 4 times a day
  Other Names: Moxifloxacin Hydrochloride 5mg/mL + Dexamethasone Disodium Phosphate 1mg/mL
  Arms: Vigadexa®

SUMMARY:
The purpose of this study is to evaluate the efficacy of Saturno II association on the control of ocular inflammation post-phacoemulsification

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes, aged 18 years or more;
* Participants presenting the diagnosis of cataract with indication for surgery by the phacoemulsification procedure;
* Participants who undergo surgery in only 1 eye at a time;
* Participants with intraocular pressure (IOP) ≤ 20 mmHg;
* Signed consent.

Exclusion Criteria:

* Used non-steroidal anti-inflammatory drugs or topical steroids or systemic inhalers within 21 days prior to randomization of the clinical trial;
* Performing the surgery for the second time, to correct the previous procedure or to change the lens;
* Decompensated glaucoma or ocular hypertension with IOP above 21 mmHg;
* Active ocular infectious diseases;
* History hypersensitivity to the active ingredients used in the study;
* Pregnancy or risk of pregnancy and lactating patients;
* History alcohol abuse or illicit drug use;
* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Participation in clinical trial in the year prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Control of ocular inflammation post-phacoemulsification as evaluated though the presence of cells in the anterior chamber | 16 days
  The inflammation will be evaluated though the presence of cells in the anterior chamber. For this, the number of cells per high-power field in the anterior chamber was counted and recorded on a scale where 0 indicates ≤ 5 cells, 1 = 5 to 10 cells, 2 = 11 to 20 cells, 3 = 21 to 50 cells, and 4 corresponds to ≥ 50 cells.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study | 26 days

CONTACTS AND LOCATIONS:
Locations (1):
- Allegisa, Campinas, São Paulo, Brazil